CLINICAL TRIAL: NCT02980185
Title: Laparoscopy for Primary Cytoreductive Surgery in Advanced Ovarian Cancer: a Prospective Validation and Comparison With Open Surgery.
Brief Title: Laparoscopy for Primary Cytoreductive Surgery in Advanced Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Stefano Uccella, Doctor, Università degli Studi dell'Insubria
Other Study IDs: 541
Record Dates: First submitted 2016-11-26; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Residual Tumor; Disease-free Survival; Overall Survival
MeSH Terms: conditions — Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Laparoscopic primary cytoreduction: Patients in whom primary cytoreduction was performed using a laparoscopic approach
  Interventions: Procedure: Laparoscopic primary cytoreduction
- Abdominal primary cytoreduction: Patients in whom primary cytoreduction was performed using an open abdominal approach

INTERVENTIONS:
Procedure: Laparoscopic primary cytoreduction — Primary cytoreduction for ovarian cancer performed through a completely minimally-invasive approach
  Groups: Laparoscopic primary cytoreduction

SUMMARY:
To assess the feasibility, Residual Tumor, complication rate and survival of totally laparoscopic primary cytoreduction in carefully selected patients with Advanced Ovarian Cancer, compared with abdominal primary cytoreduction in a single-Institution, single-surgeon prospective series.

DETAILED DESCRIPTION:
All patients with presumed stage III-IV ovarian cancer and clinical conditions allowing aggressive surgery were candidate to possible primary cytoreduction with the aim of achieving residual tumor=0. A definite protocol was adopted: after radiological preoperative evaluation with PET-CT scan, all patients underwent laparoscopic evaluation with the Fagotti score. Once considered suitable for primary debulking surgery, the possibility of attempting laparoscopic cytoreduction was carefully evaluated using strict selection criteria; patients were divided in two groups, based on the type of surgical approach. At the end of laparoscopic primary cytoreduction, a ultra-low pubic minilaparotomy was performed to extract surgical specimens and to perform laparoscopic hand-assisted exploration of the abdominal organs, in order to ensure complete excision of the disease. Surgical data, optimal cytoreduction (defined as residual tumor=0) rates and survival outcomes were investigated.

ELIGIBILITY:
Inclusion Criteria:

* Primary Ovarian cancer
* Epithelial histotype
* Stage III-IV disease

Exclusion Criteria:

* Anesthesiological contraindication to primary cytoreduction
* Extension of disease contraindicating primary cytoreduction

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing primary cytoreduction for stage III-IV ovarian cancer at the Sacred Heart Hospital, Negrar, Italy
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2007-06; Primary Completion 2015-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Residual tumor at the end of surgery (using the completeness of cytoreduction score) | June 2007 - July 2015

SECONDARY OUTCOMES:
Disease-free Survival | June 2007 - July 2016
Overall Survival | June 2007 - July 2016

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Uccella, MD, PhD, Study Chair — Università degli Studi dell'Insubria
Locations (1):
- Department of Obstetrics and Gynecology Universita' Dell'Insubria, Varese, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nezhat FR, DeNoble SM, Liu CS, Cho JE, Brown DN, Chuang L, Gretz H, Saharia P. The safety and efficacy of laparoscopic surgical staging and debulking of apparent advanced stage ovarian, fallopian tube, and primary peritoneal cancers. JSLS. 2010 Apr-Jun;14(2):155-68. doi: 10.4293/108680810X12785289143990. PMID 20932362
- [Derived] Ceccaroni M, Roviglione G, Bruni F, Clarizia R, Ruffo G, Salgarello M, Peiretti M, Uccella S. Laparoscopy for primary cytoreduction with multivisceral resections in advanced ovarian cancer: prospective validation. "The times they are a-changin"? Surg Endosc. 2018 Apr;32(4):2026-2037. doi: 10.1007/s00464-017-5899-9. Epub 2017 Oct 19. PMID 29052073